CLINICAL TRIAL: NCT03907241
Title: Title for SCGAM-03: CLINICAL PHASE III STUDY TO MONITOR THE SAFETY, TOLERABILITY AND EFFICACY OF SUBCUTANEOUS HUMAN IMMUNOGLOBULIN (OCTANORM) IN PATIENTS WITH PRIMARY IMMUNODEFICIENCY DISEASES WHO HAVE COMPLETED THE SCGAM-01 TRIAL Title for SCGAM-03 in Canada: CLINICAL PHASE III STUDY TO MONITOR THE SAFETY, TOLERABILITY AND EFFICACY OF SUBCUTANEOUS HUMAN IMMUNOGLOBULIN (OCTANORM) IN PATIENTS WITH PRIMARY IMMUNODEFICIENCY DISEASES, INCLUDING (BUT NOT LIMITED TO) THOSE WHO HAVE COMPLETED THE SCGAM-01 TRIAL
Brief Title: CLINICAL PHASE III STUDY TO MONITOR THE SAFETY, TOLERABILITY AND EFFICACY OF SUBCUTANEOUS HUMAN IMMUNOGLOBULIN (OCTANORM) IN PATIENTS WITH PRIMARY IMMUNODEFICIENCY DISEASES, INCLUDING (BUT NOT LIMITED TO) THOSE WHO HAVE COMPLETED THE SCGAM-01 TRIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCGAM-03 -; NCT02627300 (obsolete NCT alias)
Record Dates: First submitted 2018-12-07; First posted 2019-04-08 (Actual); Results first posted 2020-09-22 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Octanorm 16.5% (Experimental): octanorm 16.5%, human normal immunoglobulin for subcutaneous (SC) administration.
  Interventions: Drug: Octanorm 16.5%

INTERVENTIONS:
Drug: Octanorm 16.5% — Human normal immunoglobulin

SUMMARY:
Summary for SCGAM-03: Clinical phase III study to monitor the safety, tolerability and efficacy of subcutaneous human immunoglobulin (Octanorm) in patients with primary immunodeficiency diseases who have completed the SCGAM-01 trial.

Summary for SCGAM-03 in Canada: Clinical phase III study to monitor the safety, tolerability and efficacy of subcutaneous human immunoglobulin (octanorm) in patients with primary immunodeficiency diseases, including (but not limited to) those who have completed the SCGAM-01 trial

ELIGIBILITY:
Inclusion Criteria for SCGAM-03:

1. Completion of the main study SCGAM-01, with good tolerance of Octanorm (as determined by the investigator).
2. For adult patients: freely given written informed consent. For patients below the legal age of majority: freely given written informed consent from parents/legal guardians and written informed assent from the child/adolescent in accordance with local requirements.
3. For female patients of child-bearing potential, a negative result in a urine pregnancy test conducted at the Screening visit.
4. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Inclusion Criteria for SCGAM-03 in Canada:

Either:

SCGAM-01 patients (United States, Canada):

1. Completion of the main study SCGAM-01, with good tolerance of octanorm (as determined by the investigator).

Or:

De novo patients (Canada only):

1. C-a Age of ≥18 years and ≤75 years.

1C-b Confirmed diagnosis of PI as defined by ESID and PAGID and requiring immunoglobulin replacement therapy due to hypogammaglobulinaemia or agammaglobulinaemia. The exact type of PI should be recorded.

1. C-c Availability of the IgG trough levels of 2 previous SCIG infusions before enrolment, and maintenance of ≥5.0 g/L in the trough levels of these 2 previous infusions.

And:

2. For adult patients: freely given written informed consent. For patients below the legal age of majority: freely given written informed consent from parents/legal guardians and written informed assent from the child/adolescent in accordance with local requirements.

3. For female patients of child-bearing potential, a negative result in a urine pregnancy test conducted at the Screening Visit.

4. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Exclusion Criteria for SCGAM-03:

1. Subject being without any IgG treatment for period greater than approximately 5 weeks between the last infusion of Octanorm in the SCGAM-01 study and the first infusion of Octanorm in the SCGAM-03 study.
2. Exposure to blood or any blood product or derivative, other than IgG used for regular PID treatment, within the 3 months before the first infusion in this study.
3. Planned pregnancy during the course of the study.

Exclusion Criteria for SCGAM-03 in Canada:

* Either:

SCGAM-01 patients (United States, Canada):

1 Subject being without any IgG treatment for period greater than 5 weeks between the last infusion of octanorm in the SCGAM-01 study and the first infusion of octanorm in the SCGAM-03 study.

Or:

De novo patients (Canada only):

1C-a Acute infection requiring intravenous antibiotic treatment within 2 weeks prior to and during the screening period.

1C-b Known history of adverse reactions to IgA in other products.

1C-c Patients with body mass index >40 kg/m2.

1C-d Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products, or any component of the investigational product (such as Polysorbate 80).

1C-e Requirement of any routine premedication for IgG administration.

1C-f History of malignancies of lymphoid cells and immunodeficiency with lymphoma.

1C-g Severe liver function impairment (ALAT 3 times above upper limit of normal).

1C-h Known protein-losing enteropathies or proteinuria.

1C-i Presence of renal function impairment (creatinine >120 μM/L or creatinine >1.35 mg/dL), or predisposition for acute renal failure (e.g., any degree of pre-existing renal insufficiency or routine treatment with known nephritic drugs).

1C-j Treatment with oral or parenteral steroids for ≥30 days or when given intermittently or as bolus at daily doses ≥0.15 mg/kg.

1C-k Treatment with immunosuppressive or immunomodulatory drugs.

1C-l Live viral vaccination (such as measles, rubella, mumps and varicella) within the last 2 months prior to first infusion of octanorm.

And:

2. Exposure to blood or any blood product or plasma derivatives, other than SCIG used for regular PID treatment, within the 3 months before the first infusion of octanorm in this study.

3. Pregnant or nursing women or planned pregnancy during the course of the study.

4. Treatment with any investigational medicinal product (other than that of SCGAM-01) within 3 months prior to first infusion of octanorm.

5. Presence of any condition, that is likely to interfere with the evaluation of study medication or satisfactory conduct of the trial.

6. Known or suspected to abuse alcohol, drugs, psychotropic agents or other chemicals within the past 12 months prior to first infusion of octanorm.

7. Known or suspected HIV, HCV, or HBV infection.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Octapharma Research Site, Irvine, California
  - Octapharma Research Site, San Diego, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Papillion, Nebraska
  - Octapharma Research Site, Toledo, Ohio
  - Octapharma Research Site, Frisco, Texas
- Octapharma Research Site, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octanorm 16.5%
Started | 27
Completed | 23
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Age >=2 to <6; Age >=6 to <12; Age >=12 to <17; Age >=17 to <=75: Octanorm 16.5%
- Total: Total of all reporting groups
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75 | Total
Number analyzed (Participants) | 2 | 4 | 4 | 17 | 27
Age, Continuous [Median (Full Range); unit: years] — Patients remained in the age strata they were assigned for analysis in Study SCGAM-01 (irrespective of whether their age changed such as to imply a change of age stratum).
  years | 6.50 [6.0 to 7.0] | 9.00 [7.0 to 11.0] | 14.25 [13.0 to 15.0] | 56.12 [25.0 to 73.0] | 39.26 [6.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 13 | 17
  Male | 2 | 2 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 4 | 17 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 4 | 4 | 15 | 25
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
ABO Rhesus Blood Type [Count of Participants; unit: Participants]
  A Blood Type | 1 | 2 | 2 | 8 | 13
  AB Blood Type | 0 | 0 | 1 | 1 | 2
  O Blood Type | 1 | 2 | 1 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of All Treatment-emergent Adverse Events (TEAEs)
Description: Number of TEAEs
Time Frame: From study start to end, up to 3.5 years
Measure: Number; unit: events
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
events
  TEAEs excluding infections | 8 | 19 | 22 | 155
  Infections | 8 | 12 | 22 | 77

2. Primary Outcome: Occurrence of Temporally Associated TEAEs
Time Frame: From study start to end, up to 3.5 years
Measure: Number; unit: events
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
events
  Temporally Associated TEAEs excluding infections | 2 | 7 | 13 | 72
  Temporally Associated Infections | 5 | 6 | 11 | 45

3. Primary Outcome: Number of Temporally Associated TEAEs by Infusion Rate
Description: Number of temporally associated TEAEs by infusion rate. Only includes systemic TEAEs without infections and without infusion site reactions
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Units; unit: infusions
Units Other Than Participants: infusions
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Number analyzed (infusions) | 2 | 7 | 13 | 72
infusions
  missing | 0 | 0 | 0 | 1
  10 to <20ml/h | 1 | 0 | 0 | 0
  20 to <30ml/hr | 1 | 1 | 0 | 0
  30 to <40ml/hr | 0 | 6 | 0 | 6
  40 to <50ml/hr | 0 | 0 | 9 | 28
  50 to <60ml/hr | 0 | 0 | 4 | 3
  60 to <70ml/hr | 0 | 0 | 0 | 2
  70 to <80ml/hr | 0 | 0 | 0 | 4
  80 to <90ml/hr | 0 | 0 | 0 | 6
  90 to <100ml/hr | 0 | 0 | 0 | 22

4. Primary Outcome: Local Injection-site Reactions
Time Frame: From study start to end, up to 3.5 years
Measure: Number; unit: infusion site reactions
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
infusion site reactions | 0 | 4 | 3 | 5

5. Primary Outcome: Blood Pressure
Description: Systolic and diastolic.
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
mmHg
  Systolic Blood Pressure at Screening | 100.00 (2.828) | 105.00 (7.789) | 116.60 (6.758) | 126.21 (15.817)
  Systolic Blood Pressure End of Study | 102.50 (0.707) | 103.00 (12.302) | 114.00 (16.104) | 127.24 (12.553)
  Diastolic Blood Pressure at Screening | 63.00 (11.314) | 62.25 (6.551) | 68.50 (2.380) | 78.79 (9.407)
  Diastolic Blood Pressure at End of Study | 58.50 (13.435) | 63.75 (6.702) | 70.25 (12.842) | 73.71 (8.130)

6. Primary Outcome: Body Temperature
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 14
degrees Celsius
  Temperature at Screening | 36.85 (0.071) | 36.98 (0.287) | 36.63 (0.359) | 36.56 (0.298)
  Temperature at End of Study | 36.55 (0.354) | 36.58 (0.377) | 36.65 (0.129) | 36.57 (0.355)

7. Primary Outcome: Respiratory Rate
Time Frame: From study start to end, up to 3.5 years
Population: Not all recorded
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
breaths/minute
  Respiratory Rate at Screening | 23.50 (6.364) | 19.00 (3.830) | 16.00 (0.000) | 16.07 (2.129)
  Respiratory Rate at End of Study | 17.50 (2.121) | 15.50 (1.000) | 17.75 (2.630) | 16.47 (2.625)

8. Primary Outcome: Sodium
Description: Changes in sodium levels from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Population: Not all assessed during visits
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
mmol/L | 0.50 (0.707) | 0.25 (1.258) | 1.75 (2.217) | 0.41 (2.238)

9. Primary Outcome: Potassium
Description: Changes in potassium levels from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
mmol/L | 0.35 (0.354) | 0.25 (0.300) | 0.18 (0.340) | -0.05 (0.726)

10. Primary Outcome: Blood Glucose
Description: Changes in blood glucose from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
mmol/L | -1.03 (1.766) | 3.49 (9.017) | 0.22 (0.371) | -0.69 (1.672)

11. Primary Outcome: ALAT
Description: Changes in ALAT (alanine transaminase) from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
U/L | -2.50 (2.121) | -5.75 (8.016) | -1.50 (16.135) | 0.71 (4.074)

12. Primary Outcome: ASAT
Description: Changes in ASAT (aspartate aminotransferase) from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
U/L | -3.00 (7.071) | -4.00 (5.354) | -3.00 (11.633) | 0.59 (5.885)

13. Primary Outcome: LDH
Description: Changes in LDH (lactate dehydrogenase) from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
U/L | 23.50 (60.104) | -110.50 (131.751) | -52.50 (41.348) | -8.47 (26.779)

14. Primary Outcome: Total Bilirubin
Description: Changes in total bilirubin from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
umol/L | 0.86 (1.209) | 0.94 (1.095) | 1.58 (2.309) | 0.52 (2.793)

15. Primary Outcome: Blood Urea Nitrogen
Description: Changes in blood urea nitrogen from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 11
mmol/L | 0.36 (1.010) | -2.12 (3.124) | 0.09 (1.468) | -0.49 (1.154)

16. Primary Outcome: Creatinine
Description: Changes in creatinine from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
umol/L | -4.86 (5.626) | -27.72 (54.837) | 4.20 (6.431) | -0.62 (10.959)

17. Primary Outcome: Urine pH
Description: Changes in urine pH from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 16
pH | 0.00 (1.414) | 0.13 (2.056) | -0.50 (0.913) | -0.34 (0.889)

18. Primary Outcome: Number of Participants With a Change in Urine Glucose
Description: Number of Participants with a Change in Urine Glucose
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Participants
  From Normal to Normal | 2 | 4 | 4 | 15
  From High Non-CS to Normal | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 0 | 1

19. Primary Outcome: Number of Participants With a Change in Urine Ketones
Description: Number of Participants With a Change in Urine Ketones at baseline and end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Participants
  From Normal to Normal | 2 | 4 | 4 | 13
  From Normal to High Non-CS | 0 | 0 | 0 | 1
  From High Non-CS to Normal | 0 | 0 | 0 | 2
  From High Non-CS to Missing | 0 | 0 | 0 | 1

20. Primary Outcome: Number of Participants With a Change in Urine Leukocytes
Description: Number of participants with a change in urine leukocytes at baseline and end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Participants
  From Normal to Normal | 2 | 3 | 4 | 14
  From Normal to High Non-CS | 0 | 0 | 0 | 1
  From Normal to Missing | 0 | 1 | 0 | 2

21. Primary Outcome: Number of Participants With a Change in Urine Hemoglobin
Description: Number of participants with a change in urine hemoglobin at baseline and end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Participants
  From Normal to Normal | 2 | 4 | 4 | 14
  From Normal to High Non-CS | 0 | 0 | 0 | 1
  From High Non-CS to Normal | 0 | 0 | 0 | 1
  From High Non-CS to Missing | 0 | 0 | 0 | 1

22. Primary Outcome: Complete Red Blood Cell Count
Description: Changes in complete red blood cell count from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
10^12 cells/L | 0.14 (0.311) | -0.06 (0.256) | 0.17 (0.321) | 0.01 (0.287)

23. Primary Outcome: Haematocrit
Description: Changes in haematocrit from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
L/L | 0.02 (0.034) | 0.00 (0.013) | 0.02 (0.032) | 0.00 (0.030)

24. Primary Outcome: Haemoglobin
Description: Changes in haemoglobin from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
g/L | 8.00 (7.071) | -2.08 (4.198) | 4.25 (11.673) | 1.29 (8.513)

25. Primary Outcome: Complete White Blood Cell Count
Description: Changes in complete white blood cell count from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
10^9 cells/L | 1.45 (1.626) | -0.05 (1.034) | 0.40 (1.655) | -0.24 (1.722)

26. Secondary Outcome: Measurement of Trough Total IgG Levels
Description: Measurement of trough total IgG levels from baseline to end of study
Time Frame: From study start to end, up to 3.5 years
Population: Not all collected
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
g/L
  IgG at Screening | 10.99 (2.143) | 11.92 (3.352) | 12.17 (2.731) | 13.17 (3.236)
  IgG at End of Study: number analyzed (Participants) | 2 | 4 | 4 | 16
  IgG at End of Study | 12.50 (3.048) | 15.45 (7.359) | 9.38 (1.842) | 13.28 (3.336)

27. Secondary Outcome: Number of Participants With Serious Bacterial Infections (SBIs).
Description: Number of participants with serious bacterial infections
Time Frame: From study start to end, up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 2 | 4 | 4 | 17
Participants | 0 | 0 | 0 | 1

28. Secondary Outcome: SF-36 Health Survey.
Description: Quality of Life for patients >= age 14 assessed using the Short Form 36 Health survey. Likert like scale.
  The responses given by patients were combined to create 8 SF-36 scores: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health
  36 questions that fall into 4 Sub scale scoring ranges: Score 1-5: Where 1 is more favorable than 5 Score 1-3: Where 3 is more favorable than 1 Score 1-5: Where 5 is more favorable than 1 Score 1-6: Where 1 is more favorable than 6 The raw subscale scores are converted into a scale score between 0 to 100 using the Quality Metric Health Outcomes™ Scoring Software 2.0 Scale Title of final scales is: Physical and Mental Health Component Summary Scores Range: Lowest = 0 and highest = 100 where a high score equates to a more favorable health state
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Age >=12 to <17 | Age >=17 to <=75
Number analyzed (Participants) | 1 | 17
score on a scale
  Physical Health Score | 12.39 | 0.42 (6.922)
  Mental Health Score | -1.12 | 0.38 (10.877)

29. Secondary Outcome: CHQ-PF50 (Child Health Questionnaire-Parent Form)
Description: Quality of Life for patients ages <14 years assessed using the CHQ-PF50. Measured values represent change in score from baseline to end of study.
  Two summary scores were derived: physical and psychosocial. In accord with the scoring manual, computed scores were transformed giving each scale a possible range from 0 to 100, with the exception of change in health, with a possible range from 1 to 5. For all CHQ-PF50 scales, higher scores indicated more positive functioning or better health status.
Time Frame: From study start to end, up to 3.5 years
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age >=2 to <6: Age >=2 to <6
- Age >=6 to <12: Age >=6 to <12
- Age >=12 to <17: Age >=12 to <17
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17
Number analyzed (Participants) | 2 | 3 | 2
score on a scale
  Physical Summary Score | -0.79 (5.032) | 0.94 (6.800) | 2.76 (2.683)
  Psychosocial Summary | -9.07 (12.361) | 0.50 (2.679) | 9.92 (20.860)

ADVERSE EVENTS:
Time Frame: From study start to end, up to 3.5 years
Arm/Group | Age >=2 to <6 | Age >=6 to <12 | Age >=12 to <17 | Age >=17 to <=75
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/4 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 2/4 | 4/17
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 4/4 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age >=2 to <6 (N=2) | Age >=6 to <12 (N=4) | Age >=12 to <17 (N=4) | Age >=17 to <=75 (N=17)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age >=2 to <6 (N=2) | Age >=6 to <12 (N=4) | Age >=12 to <17 (N=4) | Age >=17 to <=75 (N=17)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Oedema (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal infiltrates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dypsnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interverterbral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood alcohol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postmenopause (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (4)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (2) | 2 (3) | 3 (3)
Infusion site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (8)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (6) | 8 (29)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: US and Canada (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT03907241/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03907241/SAP_003.pdf
  • Study Protocol: US only (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03907241/Prot_004.pdf